CLINICAL TRIAL: NCT06467019
Title: Impact of an Interactive and Informative Exhibition on Benzodiazepine Use on Deprescription.
Brief Title: Informative Exhibition for Deprescribing Benzodiazepines
Acronym: ESUB
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-59
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Benzodiazepine-Related Disorders
Keywords: Benzodiazepines; Deprescriptions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before intervention: This group will consist of patients who attended the primary care center before the implementation of the intervention.
- After intervention: This group will consist of patients who will attend the primary care center after the implementation of the intervention.
  Interventions: Other: Informative Session

INTERVENTIONS:
Other: Informative Session — The intervention consists of implementing an interactive exhibition on the risks of chronic benzodiazepine treatment in the waiting room of a primary care center. Additionally, the health professionals at the center will receive a single informative session on the same topic.
  Groups: After intervention

SUMMARY:
The goal of this trial is to determine if an interactive and informative exhibition in the waiting room of a Primary Care Clinic can reduce the use of benzodiazepines in adults. The main question it aims to answer is:

• Does an interactive and informative exhibition reduce the number of participants using benzodiazepines? Researchers will compare benzodiazepine consumption before and after the interactive and informative exhibition implementation at study center.

Participants will receive an informative and interactive exhibition on the risks of chronic benzodiazepine use. A single informative session on the same topic will be conducted for health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 99 years of age.
* Attended at the Baix-a-Mar Primary Care Center during the study period.

Exclusion Criteria:

* Severe mental health disease
* Displaced patients or those who do not have an assigned doctor at the center.
* Participation in another study involving an experimental intervention during the period of the present study that affects benzodiazepine prescription.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community population assigned to a primary care center.
Sampling Method: Non-Probability Sample
Enrollment: 6410 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Chronic treatment with benzodiazepines | 1 year
  Percentage of patients treated chronically with benzodiazepines, based on electronic prescription data.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Milozzi, MD, Principal Investigator — Centro de Salud Vilanova i la Geltrú 3 Baix A Mar-CSAPG
Locations (1):
- Centro de Salud Vilanova i la Geltrú 3 Baix A Mar, Vilanova i la Geltrú, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.